CLINICAL TRIAL: NCT06588140
Title: Comparison of Retention Between Different Duplication Techniques of Complete Dentures: Conventional Versus CAD/CAM: A Within Subject Controlled Clinical Trial
Brief Title: Conventional Versus 3D Printing Duplication Techniques of Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M. Refai, Lecturer of Oral and Maxillofacial Prosthodontics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FDASU-Rec IR032421
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Denture,Complete; Edentulous Alveolar Ridge
Keywords: CAD-CAM; Complete Dentures; Copying , Denture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional heat-cured duplication technique. (Active Comparator): Duplication of refitted complete removable dentures by conventional heat-cured technique from heat-cured polymethyl methacrylate resin.
  Interventions: Device: Duplicated refitted complete denture made from conventionally heat-cured polymethyl methacrylate.
- 3d Printed CAD/CAM duplication technique from Pink polymethyl methacrylate base resin (Experimental): Duplication of a refitted complete removable denture will be produced using a 3D-printed CAD/CAM technique where the denture base will be printed separately using pink base polymethyl methacrylate resin, and the teeth will be printed as one unit using tooth-colored resin, followed by assembling the two components.
  Interventions: Device: Duplicated refitted complete denture made from 3D-printed CAD/CAM pink polymethylmethacrylate acrylic resin.
- 3d Printed CAD/CAM duplication technique from white polymethyl methacrylate base resin (Experimental): Duplication of a refitted complete removable denture will be produced using a 3D-printed CAD/CAM technique where the denture will be printed as a single unit using tooth-colored resin, and the denture flange will be veneered with pink resin.
  Interventions: Device: Duplicated refitted complete denture made from 3D-printed CAD/CAM white polymethylmethacrylate acrylic resin.

INTERVENTIONS:
Device: Duplicated refitted complete denture made from conventionally heat-cured polymethyl methacrylate. — The duplication of a refitted complete removable denture will be performed using conventional heat-cured polymethyl methacrylate through the conventional heat-cured polymerization technique.
  Arms: conventional heat-cured duplication technique.
Device: Duplicated refitted complete denture made from 3D-printed CAD/CAM pink polymethylmethacrylate acrylic resin. — The duplication of a refitted complete removable denture will be performed using a 3D-printed CAD/CAM technique, where the denture base is printed separately with pink polymethyl methacrylate resin, and the teeth are printed as a single unit using tooth-colored resin, followed by the assembly of the two components.
  Arms: 3d Printed CAD/CAM duplication technique from Pink polymethyl methacrylate base resin
Device: Duplicated refitted complete denture made from 3D-printed CAD/CAM white polymethylmethacrylate acrylic resin. — The duplication of a refitted complete removable denture will be performed using a 3D-printed CAD/CAM technique, where the denture base is printed as a single unit using tooth-colored resin, and the denture flange will be veneered with pink polymethyl methacrylate resin.
  Arms: 3d Printed CAD/CAM duplication technique from white polymethyl methacrylate base resin

SUMMARY:
Twenty completely edentulous patients with old, removable dentures with ill-fitting maxillary dentures, proper vertical dimension, and proper occlusion will be recruited for this trial. They will be rehabilitated with duplicated complete dentures manufactured by conventional and two different 3D-printed CAD-CAM Complete Removable Dentures techniques.

Outcomes will be evaluated, including denture retention, which will be evaluated using a digital force gauge, and occlusal force distribution by using a t-scan.

DETAILED DESCRIPTION:
The study will be conducted at the outpatient clinic of the Oral and Maxillofacial Prosthodontics Department, Faculty of Dentistry, Ain Shams University. This within-subject controlled clinical trial will involve twenty completely edentulous patients with old, ill-fitting maxillary complete dentures, who will be selected and recruited following approval by the Research Ethics Committee of the Faculty of Dentistry, Ain Shams University (FDASU-REC). These patients will be rehabilitated with duplicated complete dentures produced through conventional methods and two distinct 3D-printed CAD/CAM techniques.

Group I: The duplication of a refitted complete removable denture will be performed using the conventional heat-cured technique.

Group II: The refitted complete denture will be duplicated using a 3D-printed CAD/CAM technique, where the denture base will be printed separately with pink resin, and the teeth will be printed as a single unit in tooth-colored resin, followed by assembly of the two components.

Group III: The refitted complete denture will be duplicated using a 3D-printed CAD/CAM technique, with the entire denture printed as a single unit in tooth-colored resin, and the denture flange veneered with pink resin.

Outcomes will be evaluated by measuring denture retention with a digital force gauge and occlusal force distribution using the T-Scan system. The collected data will be recorded, tabulated, and subjected to statistical analysis using appropriate tests for group comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with old complete dentures without lost vertical dimension.
2. Patients with correct centric occluding relation.
3. The dentures should be esthetically and functionally satisfactory and exhibit reasonable retention and stability

Exclusion Criteria:

1. The presence of ridge or soft tissue pathology.
2. Diminished saliva production.
3. A history of medications affecting saliva quantity or quality.
4. Patients with temporomandibular joint problems.
5. The presence of sever ridge undercut.
6. Debilitated patients

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Retention of maxillary complete denture | at the time of denture insertion
  The retention of a maxillary complete denture will be assessed using a digital force gauge meter, with retention measurements recorded in Newtons.

SECONDARY OUTCOMES:
Evaluation of occlusal force distribution between right and left side | at the time of denture insertion
  Occlusal force distribution will be assessed using the T-Scan III, with the results expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Amany M Saad Farahat, PHD, Principal Investigator — Ain Shams Univeristy; Yasmine S Elsherbeeny, PHD, Principal Investigator — Ain Shams Univeristy
Locations (1):
- Ain Shams University, Cairo, Egypt